CLINICAL TRIAL: NCT06290973
Title: Quality of Life and Health Perception After Surgery of Varicose Veins
Status: Completed | Type: Observational
Sponsor: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Principal Investigator, Diana Gutierrez Castillo, PhD, Hospital Clínico Universitario de Valladolid
Other Study IDs: PI-23-3017
Record Dates: First submitted 2023-11-23; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Quality of Life; Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgery of varicose veins — including ablation with radiofrequency, phlebectomy and saphenectomy.

SUMMARY:
The aim of this study is to analyze changes in health perception and quality of life in patients after surgery for varicose veins using clinical score VCSS and QoL scores SF12 as general health questionary and Veines QoL/Sym as disease specific questionary.

ELIGIBILITY:
Inclusion Criteria:

* patients with reflux in saphenous vein

Exclusion Criteria:

* no reflux in saphenous vein

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with varicose veins undergoing surgery between january and february of 2023 in Valladolid Clinical Hospital
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
changes in qol questionarie SF-12 after surgery of varicose veins | before and 90 days after surgery
  measured in SF-12 score
changes in qol questionarie Veines QoL/Sym after surgery of | before and 90 days after surgery
  measured in Veines Qol/Sym score

SECONDARY OUTCOMES:
changes in VCSS after surgery of varicose veins | before and 90 days after surgery
  measured in VCSS score

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital CLínico Universitario de Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No